CLINICAL TRIAL: NCT07064486
Title: A Phase 3, Randomized, Open Label Trial Comparing Efficacy and Safety of BGM0504 Versus Semaglutide Once Weekly as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: A Study of BGM0504 in Participants With Type 2 Diabetes in Indonesia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGM0504-Ⅲ-T2DM-02-IDN
Record Dates: First submitted 2025-07-11; First posted 2025-07-14 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5 mg BGM0504 (Experimental): 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
  Interventions: Drug: BGM0504
- 10 mg BGM0504 (Experimental): 10 mg BGM0504 administered SC once a week.
  Interventions: Drug: BGM0504
- 1 mg Semaglutide (Active Comparator): 1 mg semaglutide administered SC once a week
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: BGM0504 — Administered SC
  Arms: 5 mg BGM0504
Drug: BGM0504 — Administered SC
  Arms: 10 mg BGM0504
Drug: Semaglutide — Administered SC
  Arms: 1 mg Semaglutide

SUMMARY:
This trial is conducted in Indonesia. The aim of the trial is to evaluate the efficacy and safety of BGM0504 versus semaglutide as add-on to metformin in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* ○ Have been diagnosed with type 2 diabetes mellitus (T2DM);

  * Be on stable treatment with unchanged dose of metformin ≥1500 mg/day or <1500 mg/day but ≥1000 mg/day (the maximum tolerated dose) for at least 8 weeks prior to screening
  * Have a BMI ≥23 kilograms per meter squared (kg/m²) at screening;
  * Be of stable weight (± 5%) for at least 3 months before screening;
  * Have HbA1c between ≥7.5% and ≤11.0% at screening

Exclusion Criteria:

* ○ Previous diagnosis of type 1 diabetes, special type diabetes;

  * Have suffered the malignancy within the past 5 years (except cured basal cell carcinoma of the skin, cervical carcinoma in situ), or being evaluated for an underlying malignancy;
  * Have the acute or chronic pancreatitis;
  * Known to be allergic to 3 or more kinds of foods or medications, or allergic to GLP-1 agonist or metformin, or have a severe allergic disease (asthma, urticaria, eczematous dermatitis, etc.) at screening;
  * Have a serious mental illness or speech impediment and be unable to fully understand the study;
  * Suspected or confirmed history of alcohol or drug abuse;
  * Have had a history of ≥2 severe hypoglycemic episodes in the past 1 year;
  * Other conditions that may impact the assessment of investigational products, as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 24
  Change from baseline in HbA1c after 24 weeks of treatment.

SECONDARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 12
  Change from baseline in HbA1c after 12 weeks of treatment.
Change From Baseline in Body Weight | Week 0 to Week 24
  Change from baseline in body weight after 24 weeks of treatment.
Percentage of Participants With HbA1c Target Value of <7% | Week 0 to Week 24
  Percentage of Participants With HbA1c Target Value of <7% after 24 weeks of treatment.
Percentage of Participants With HbA1c Target Value of <5.7% | Week 0 to Week 24
  Percentage of Participants With HbA1c Target Value of <5.7%after 24 weeks of treatment.
Change From Baseline in Fasting Serum Glucose | Week 0 to Week 24
  Change from baseline in FPG after 24 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Indonesia (4):
  - RS Universitas Indonesia, Depok, West Java
  - RSUP Fatmawati, Jakarta
  - RSUP Persahabatan, Jakarta
  - RSUPN Dr. Cipto Mangunkusumo, Jakarta